CLINICAL TRIAL: NCT00393445
Title: Effect of GLP-1 on Glucose Metabolism in Healthy Subjects and Patients With T2DM. Part 1: A Pilot Study to Assess the Efficacy of Exendin(9-39)Amide as a GLP-1 Receptor Antagonist in Healthy Subjects
Brief Title: Exendin(9-39)Amide as a Glucagon-like Peptide-1 (GLP-1) Receptor Antagonist in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Research Foundation (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joerg Schirra, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: DOF-Ex; DFG Schi 527/1-2
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Hyperglycemia
Keywords: GLP-1; Exendin(9-39); Insulin; Glucagon; Human physiology
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — glucagon-like peptide 1 (7-36)amide; Glucagon-Like Peptide 1; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous infusion (Experimental): intravenous infusion of test substances
  Interventions: Drug: GLP-1 control; Drug: GLP-1 and Exendin(9-39) 300; Drug: saline control; Drug: GLP-1 and Exendin(9-39) 600; Drug: GLP-1 and Exendin(9-39) 900; Drug: GLP-1 and Exendin(9-39) 1200

INTERVENTIONS:
Drug: GLP-1 control — intravenous infusion of GLP-1
  Other Names: GLP-1(7-36)amide
Drug: GLP-1 and Exendin(9-39) 300 — intravenous infusion of exendin(9-39) at 300 pmol/kg/min during GLP-1 at 0.3 and 0.9 pmol/kg/min
Drug: saline control — intravenous infusion of saline
Drug: GLP-1 and Exendin(9-39) 600 — intravenous infusion of exendin(9-39) at 600 pmol/kg/min during GLP-1 at 0.3 and 0.9 pmol/kg/min
Drug: GLP-1 and Exendin(9-39) 900 — intravenous infusion of exendin(9-39) at 900 pmol/kg/min during GLP-1 at 0.3 and 0.9 pmol/kg/min
Drug: GLP-1 and Exendin(9-39) 1200 — intravenous infusion of exendin(9-39) at 1200 pmol/kg/min during GLP-1 at 0.3 and 0.9 pmol/kg/min

SUMMARY:
The purpose of this study is to determine the dose of the GLP-1 receptor antagonist exendin(9-39) which blocks the insulinotropic action of synthetic GLP-1 by at least 95%.

DETAILED DESCRIPTION:
Following a meal, gut-produced incretin hormones such as glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) are released into the circulation. GLP-1 and GIP, the two dominant incretin hormones, are part of a natural endogenous system involved in maintaining glucose homeostasis. In the presence of normal or elevated, but not low, glucose concentration, both GLP-1 and GIP increase insulin secretion from pancreatic islet beta-cells (β-cells). GLP-1 also lowers glucagon secretion from pancreatic alpha-cells and delays nutrient delivery from the stomach by inhibiting gastric emptying. This rise in insulin concentration enhances glucose clearance in peripheral tissues such as muscle, and the lower glucagon concentration combined with the rise in insulin reduces hepatic glucose production. By enhancing glucose clearance and lowering hepatic glucose production, the post-meal glucose excursion is reduced.

However, the role that each incretin has in glucoregulation is not fully understood. Use of a GLP-1 antagonist, exendin (9-39)NH2, will allow for the assessment of non-GLP-1 incretin's role in glucoregulation. Therefore, it is of great interest to examine the role that specific incretins have in glucoregulation in patients with T2DM.

Exendin(9-39) has been shown a specific and reversible antagonist at the human GLP-1 receptor in vivo. In initial validation studies intravenous exendin(9-39) dose-dependently reduced the insulinotropic action of intravenous GLP-1. The maximal dose of 300 pmol/kg/min used in these studies was sufficient to reduce GLP-1 stimulated insulin plasma levels by about 83%. However, to quantify the contribution of incretin hormones to the incretin effect as stated above a nearly complete inhibition of the GLP-1 action is necessary.

Therefore the purpose of this pilot study is to characterize the dose-response characteristics of exendin(9-39) more completely and to find a dosage which inhibits the insulinotropic action of GLP-1 by at least 95%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (postmenopausal, surgically sterile or using double-barrier method of contraception) healthy volunteers
* Age 18-65 years
* Hemoglobin A1c (HbA1c) < 6%
* Body mass index (BMI) < 30 kg/m2
* Must have a fasting blood glucose below 100 mg/dl at screening and on all study days
* Able to provide written informed consent prior to study participation
* Able to communicate well with the investigator and comply with the requirements of the study

Exclusion Criteria:

* Diabetes mellitus
* Fasting triglycerides > 5.1 mmol/L (> 450 mg/dL) within the past 4 weeks.
* Treatment with systemic steroids and thyroid hormone
* Patients with any history of gastrointestinal surgery, e.g. partial bowel resections, partial gastric resections, etc.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Past medical history of clinically significant electrocardiogram (ECG) abnormalities or a family history of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study. The investigator should be guided by evidence of any of the following:

  * history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
  * history or clinical evidence of pancreatic injury or pancreatitis
  * history or presence of impaired renal function as indicated by abnormal creatinine or urea values or abnormal urinary constituents (e.g., albuminuria)
  * evidence of urinary obstruction or difficulty in voiding at screening
* Polymorphonuclears < 1500/µL at inclusion or platelet count < 100,000/μL at screening and baseline.
* Evidence of liver disease as indicated by abnormal liver function tests such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-11; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To assess the effect of increasing doses of exendin(9-39) on first and second phase insulin secretion stimulated by intravenous GLP-1 during hyperglycemia | within the actual study period

SECONDARY OUTCOMES:
To assess the effect of increasing doses of exendin(9-39) on plasma glucagon levels decreased by intravenous GLP-1 during hyperglycemia | within the actual study period

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, MD, Study Chair — Clinical Research Unit (CRU), Department of Internal Medicine II-Grosshadern, Ludwig-Maximilans-University of Munich
Locations (1):
- Ludwig Maximilians University, Clinical Research Unit, Munich, Germany

REFERENCES:
- [Result] Schirra J, Sturm K, Leicht P, Arnold R, Goke B, Katschinski M. Exendin(9-39)amide is an antagonist of glucagon-like peptide-1(7-36)amide in humans. J Clin Invest. 1998 Apr 1;101(7):1421-30. doi: 10.1172/JCI1349. PMID 9525985
- [Result] Schirra J, Katschinski M, Weidmann C, Schafer T, Wank U, Arnold R, Goke B. Gastric emptying and release of incretin hormones after glucose ingestion in humans. J Clin Invest. 1996 Jan 1;97(1):92-103. doi: 10.1172/JCI118411. PMID 8550855